CLINICAL TRIAL: NCT01436435
Title: Jetstream NAVITUS™ System Endovascular Therapy Post-market Registry (JET)
Brief Title: The Jetstream (JET) Post-market Registry
Acronym: JET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1465
Record Dates: First submitted 2011-09-02; First posted 2011-09-19 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Peripheral Arterial Diseases
Keywords: PAD; peripheral artery disease; atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Jetstream Atherectomy System (Experimental): Patients with symptomatic peripheral vascular disease undergoing percutaneous intervention including Atherectomy utilizing the Jetstream Atherectomy System with or without adjunctive therapy.
  Interventions: Device: Jetstream Atherectomy System

INTERVENTIONS:
Device: Jetstream Atherectomy System — Atherectomy

SUMMARY:
The scope of the JET registry to observe long term treatment effects of Jetstream Navitus on various lesions types/morphologies.

DETAILED DESCRIPTION:
* To observe the treatment effects of the Jetstream NAVITUS System in long, occluded, diffuse, thrombotic or calcified lesions in peripheral arterial disease of the common femoral, superficial femoral, or popliteal arteries.
* To assess and quantify vessel patency 1 year post atherectomy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age.
* The target de novo or restenotic Percutaneous Transluminal Angioplasty (PTA) lesion(s) is/are located in the common femoral, superficial femoral or popliteal arteries.
* The reference vessel lumen (proximal to target lesion) is ≥ 4.0mm.
* Evidence of ≥ 70% stenosis or occlusion confirmed by angiography.
* Guidewire must cross lesion(s) within the true lumen, without a sub-intimal course before the patient is considered as entered into the study.
* Patient is an acceptable candidate for percutaneous intervention using the Jetstream NAVITUS System in accordance with its labeled indications and instructions for use.
* Lesion length ≥ 4cm.
* Patient has a Rutherford category score of 1-3.
* Patient has signed approved informed consent.
* Patient is willing to comply with the follow-up evaluations at specified times.

Exclusion Criteria:

* Patient has an uncontrollable allergy to nitinol, stainless steel or other stent materials or to contrast agent.
* Patient is unable to take appropriate anti-platelet therapy.
* Patient has no patent distal runoff vessels.
* Patient has critical limb ischemia (i.e., Rutherford class 4-6)
* Limited vascular access that precludes safe advancement of the Jetstream NAVITUS System to the target lesion(s).
* Interventional treatment is intended for in-stent restenosis.
* Patient has target vessel with moderate or severe angulation (e.g., >30 degrees) or tortuosity at the treatment segment.
* Patient has a history of coagulopathy or hypercoagulable bleeding disorder.
* Patient is receiving hemodialysis or has significantly impaired renal function (creatinine is > 2.5 mg/dl) at the time of treatment.
* Patient has evidence of intracranial or gastrointestinal bleeding within the past 3 months.
* Patient has had severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days.
* Patient has had surgical or endovascular procedure in the same vascular territory within 30 days prior to the index procedure.
* Patient has any planned surgical intervention or endovascular procedure within 30 days after the index procedure.
* Use of another debulking device during the index procedure prior to the Jetstream NAVITUS System will exclude the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Columbia University
Locations (11):
- United States (11):
  - Nelson Bernardo MD, Washington D.C., District of Columbia
  - Robert Beasley, MD, Miami, Florida
  - Nicolas Shammas, MD, Davenport, Iowa
  - Lawrence Garcia, MD, Boston, Massachusetts
  - Vinay Kumar, Laurel, Mississippi
  - Andrey Espinoza, MD, Flemington, New Jersey
  - Sotir Polena, MD, Huntington, New York
  - Rajesh Dave, MD, Harrisburg, Pennsylvania
  - Ali Amin, MD, West Reading, Pennsylvania
  - Lee Butterfield, MD, Columbia, South Carolina
  - Chris Metzger, MD, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Jetstream Atherectomy System
Started | 241
Completed | 177
Not Completed | 64

BASELINE CHARACTERISTICS:
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 159
Region of Enrollment [Number; unit: participants]
  United States | 241

OUTCOME MEASURES:

1. Primary Outcome: Binary Restenosis
Description: Percentage of patients with binary restenosis at 12 months as defined by duplex ultrasound derived systolic velocity ratio >2.5. Binary restenosis will be measured by duplex ultrasound technology.
Time Frame: 12 months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 184 participants were not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 57
percentage of patients | 22.8

2. Secondary Outcome: Procedural Success
Description: Percentage of patients with successful revascularization of target vessel defined as ≤ 30% residual diameter stenosis following atherectomy +/- adjunctive therapy
Time Frame: Index Procedure
Population: Analysis was intention to treat; all participants in the study were evaluated to provide the information needed for this endpoint
Measure: Number; unit: percentage of patients
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 241
percentage of patients | 98.3

3. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: Improvement in Ankle-Brachial Index (ABI) by ≥0.10 from the pre-procedure value. ABI is a quick, non-invasive test that compares your blood pressure measured at your ankle with your blood pressure measured at your arm.
Time Frame: 30 days
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 22 participants were not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 219
percentage of patients | 73.5

4. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: as for outcome 3
Time Frame: 6 months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 51 participants were not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 190
percentage of patients | 54.7

5. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: as for outcome 3
Time Frame: 12 months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 64 participants were not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 177
percentage of patients | 58.2

6. Secondary Outcome: Major Adverse Events (MAE)
Description: Number of Major Adverse Events as defined by amputation, death, Target Lesion Revascularization, Target Vessel Revascularization, Myocardial Infarction or angiographic distal embolization that requires a separate intervention or hospitalization through 30 days
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: Major Adverse Events
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 219
Major Adverse Events | 5

ADVERSE EVENTS:
Time Frame: Index procedure through 12 month follow up
Arm/Group | Jetstream Atherectomy System
Serious Adverse Events (participants affected / at risk) | 42/241
Other Adverse Events (participants affected / at risk) | 38/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Jetstream Atherectomy System (N=241)
Target Vessel Revascularization/ Target Lesion Revascularization (Vascular disorders) | 38 (38) — Device and/or Procedure Related
Distal Embolization Requiring a Separate Intervention (Vascular disorders) | 3 (3) — Device Related
Amputation (Surgical and medical procedures) | 1 (1) — Device Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Jetstream Atherectomy System (N=241)
Peripheral Artery Disease (Vascular disorders) | 38 (49) — Includes target and non-target study limbs/lesions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No